CLINICAL TRIAL: NCT07246772
Title: Effects of Electrical Muscle Stimulation Exercise on Lower, Upper Extremity and Core Strength in Sedentary Women
Brief Title: Effects of EMS on Strength in Sedentary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra Korkmaz Salkılic, Phd, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EsraEMS2025; Ondokuz Mayıs University (Other: Ondokuz Mayıs University Clinical Research Ethics Committee (approval number: 021/482).)
Record Dates: First submitted 2025-07-24; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sedentary Lifestyle; Muscle Stimulation
Keywords: Electro muscle stimulation, strength, anthropometric, sedentary
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the electrical muscle stimulation group or the control group."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Electrical Muscle Stimulation Exercise Group (Experimental): Participants in this group received neuromuscular electrical stimulation (EMS) concurrently with a standardized exercise protocol for a duration of 20 minutes
  Interventions: Device: Electrical Muscle Stimulation (EMS)
- Exercise-Only Group (Active Comparator): A standardized exercise protocol performed for 20 minutes without the use of EMS
  Interventions: Behavioral: Standard Exercise Protocol

INTERVENTIONS:
Device: Electrical Muscle Stimulation (EMS) — Intervention 1: Exercise + EMS Intervention Type: Device (because EMS is applied using a device)
  Intervention Name: Electrical Muscle Stimulation (EMS)
  Description: Simultaneous electrical stimulation is applied to the lower extremity muscles using an EMS device. The application lasts for 20 minutes and is performed concurrently with the exercise protocol.
  Arms: Arm 1: Electrical Muscle Stimulation Exercise Group
Behavioral: Standard Exercise Protocol — The standard exercise protocol is applied for 20 minutes without the use of EMS. The same protocol is also applied in the EMS group.
  Arms: Exercise-Only Group

SUMMARY:
Abstract Aim of the Study: This study aimed to compare the effects of Electro Muscle Stimulation (EMS) exercise on physical performance in sedentary women.

Methods: Our study was conducted with a total of 27 sedentary women, 12 EMS, and 15 controls, aged 19-24 years. The tests administered to the participants were the Modified Push-Up Test (MPU), Hand Grip Strength Test (HS), Bent Arm Hanging Test (BAH), Single Leg Hop Tests (SLHT) [single hop for distance (SH), triple jump for distance (TH) and cross triple jump for distance (CH), medial side triple jump for distance (MSTH)], Deep squat (DS), V-Sit Flexor Test (V-sit), Sit-Up Test and Biering Sorensen (Bie-sor) tests. All tests were repeated pre-mid-post and each test period was randomized with practice cards.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the participants were determined as being between the ages of 19-24, being female, and volunteering. Exclusion criteria were those who had cardiovascular, neurological, or orthopedic disorders, were pregnant or were planning to become pregnant.

Exclusion Criteria:

Ages: 19 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Lower extremity muscle strength | Baseline, 4 weeks and 8 weeks after intervention start
  Change in lower extremity muscle strength assessed by functional performance tests at baseline, 4 weeks, and after 8 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Farivar Wellness Center, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

DOCUMENTS (3):
  • Study Protocol (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT07246772/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT07246772/SAP_001.pdf
  • Informed Consent Form (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT07246772/ICF_002.pdf